CLINICAL TRIAL: NCT05322590
Title: A Phase 1b/2 Placebo Controlled, Double Blinded Study on the Efficacy and Safety of BXQ-350 in Combination With mFOLFOX7 and Bevacizumab in Newly Diagnosed Metastatic Colorectal Carcinoma
Brief Title: BXQ-350 in Newly Diagnosed Metastatic Colorectal Carcinoma
Acronym: ASIST
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bexion Pharmaceuticals, Inc. (Industry)
Collaborators: ICON plc (Industry); CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BXQ-350.AG
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Carcinoma; Neuropathy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Enrollment will proceed in 2 stages. In the Stage 1 (open label) safety run-in phase, participants are enrolled and treated in cohorts of 3 in order to reach a maximum tolerated dose (MTD) or recommended Phase 2 Dose (RP2D). After the MTD/RP2D is established, a cohort expansion of up to 30 participants will be conducted at the RP2D. Stage 1 enrollment was completed in November 2024.
  In Stage 2, eligible participants will be randomized in a 1:1 ratio to receive either BXQ-350 at the RP2D or placebo (0.9% normal saline) intravenously (IV) administered in combination with mFOLFOX7 and bevacizumab.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 1 (open label)/Stage 2 (Randomized, Placebo controlled, Double Blind)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BXQ-350 (Experimental): BXQ-350 will be administered by IV infusion
  Interventions: Drug: BXQ-350
- Placebo (Placebo Comparator): Placebo (0.9% normal saline) will be administered by IV infusion (Stage 2 only)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BXQ-350 — BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a phospholipid located on cell membranes (clinical formulation BXQ-350). BXQ-350 will be administered by intravenous (IV) infusion over six months and continued for an additional 20 months for participants who remain eligible.
  Other Names: SapC-DOPS
  Arms: BXQ-350
Other: Placebo — Placebo will be 0.9% normal saline of matching volume to BXQ-350 administered by intravenous (IV) infusion over six months and continued for an additional 20 months for participants who remain eligible (Stage 2 only)
  Arms: Placebo

SUMMARY:
The study will assess the safety and efficacy of BXQ-350 plus modified FOLFOX7 (mFOLFOX7) and bevacizumab in participants who have newly diagnosed metastatic adenocarcinoma of the colon/rectum. The study will also evaluate if the administration of BXQ-350 with mFOLFOX7 and bevacizumab may diminish oxaliplatin induced sensory neurotoxicity, enabling participants to receive the total and planned doses of mFOLFOX7.

All participants will receive BXQ-350 by intravenous (IV) infusion along with standard of care doses of mFOLFOX and bevacizumab. The study is divided into two stages: Stage 1 will be open label and will enroll participants at increasing dose levels of BXQ-350 in order to determine the Stage 2 dose. Stage 2 will be blinded; participants will receive BXQ-350 at the established Stage 1 dose or placebo.

DETAILED DESCRIPTION:
BXQ-350 is a novel anti-neoplastic therapeutic agent configured from two components: Saposin C (SapC), an expressed (human) lysosomal protein, and the phospholipid dioleoylphosphatidyl-serine (DOPS), a cell membrane phospholipid (clinical formulation BXQ-350).Due to the presumed mechanism of action of BXQ-350, Bexion anticipates that it may have an impact on ceramides, sphingosine-1-phosphate (S1P), and inflammatory cytokine levels. In addition, pre-clinical results demonstrated that BXQ-350 induced neurite generation and protection in vitro in the PC-12 and NS20Y cell lines and significantly decreased oxaliplatin-induced cold allodynia in a model of CIPN. Thus BXQ-350 may represent a new approach to deliver a neuropathy benefit.

The unique combination of BXQ-350 along with its proven safety profile, potential efficacy, and possible neuropathy benefit makes BXQ-350 a worthwhile candidate to use in combination with standard of care treatment for mCRC to not only enhance the standard treatment of mCRC, but also to evaluate its ability to alleviate side effects related to oxaliplatin-induced sensory neurotoxicity.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet the following criteria will be considered eligible to participate in the clinical study:

1. Age ≥ 18 years of age at the time of signing the informed consent.
2. Participants have newly diagnosed Stage IV metastatic adenocarcinoma of the colon / rectum.
3. Have measurable disease at baseline based on RECIST 1.1 as determined by the local site Investigator / radiology assessment.
4. Have a life expectancy > 3 months.
5. Have ECOG Performance Status of 0 or 1.

   * Participants unable to walk because of paralysis, but who can sit without assistance/restraint and control a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
6. Have acceptable liver function defined as:

   * Total serum bilirubin ≤ 1.5 x upper limit of normal (ULN) for the study site; in participants with known Gilbert Syndrome, total bilirubin ≤ 3 x ULN, with direct bilirubin ≤ 1.5 x ULN).
   * Aspartate transaminase (AST), serum glutamic oxaloacetic transaminase (SGOT), alanine transaminase (ALT), serum glutamic pyruvic transaminase (SGPT) ≤ 3 x ULN (if liver metastases are present, then ≤ 5 x ULN is allowed).
   * Serum albumin ≥ 3 g/ dL.
7. Have acceptable renal function defined as:

   * Creatinine clearance ≥ 50 mL/minute calculated using the Cockcroft-Gault formula (Cockcroft 1976): CCr = {((140 - age) x weight kg) / (72 x SCr)} x 0.85 (if female).
   * Urine dipstick protein < 1 + (30 - 70 mg/dL), urine protein/creatinine ratio of < 1, OR 24 hour urine protein < 1g/24 hours.
8. Have acceptable bone marrow function defined as:

   * Absolute neutrophil count ≥ 1,500 cells / mm3.
   * Platelet count ≥ 100,000 cells / mm3 (unsupported, no transfusion within 7 days of enrollment).
   * Hemoglobin > 9.0 g/dL (unsupported, no transfusion within 7 days of enrollment).
9. Have acceptable coagulation parameters (anti-coagulation allowed) defined as:

   * International normalized ratio ≤ 2 x ULN unless on anticoagulation or prothrombin time within normal limits.
   * Activated partial thromboplastin time within normal limits.
10. Have a negative serum pregnancy test result at screening (females of childbearing potential [FCBP] only). Not applicable to participants who are surgically sterile (i.e., bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or who are post-menopausal. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
11. Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. FCBP whose partner(s) are non-sterilized males and non-sterilized male participants whose sexual partner(s) are FCBP must abstain from heterosexual activity or agree to use an acceptable method of contraception according to the following guidelines:

    * The reliability of sexual abstinence for male and/or female enrollment eligibility needs to be evaluated in relation to the duration of the entire period of risk associated with study interventions and the preferred and usual lifestyle of the participant. Total sexual abstinence is an acceptable method provided it is the usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or post ovulation methods), the rhythm method, and withdrawal are not acceptable methods of contraception.
    * Non-sterilized Male Participants:

      * Must use an acceptable method of contraception such as male condom plus spermicide during the entire period of risk associated with study interventions which includes the total duration of the study and the drug washout period (6 months after the last dose of study intervention) and refrain from sperm donation or banking throughout this period.
      * Vasectomized males are considered fertile and should still use a male condom plus spermicide as indicated above.
      * Even if the female partner is pregnant, male participants should still use a condom plus spermicide, as indicated above..
      * Female partners (of childbearing potential) of male participants must also use a highly effective method of contraception during the entire period of risk associated with study interventions as described above.
    * FCBP

      * Must use a highly effective method of contraception and avoid breastfeeding during the entire period of risk associated with study interventions which includes the total duration of the study and the drug washout period (9 months after the last dose of study intervention) and refrain from egg donation or banking throughout this period.
      * Non-sterilized male partners must also use a male condom plus spermicide during the entire period of risk associated with study interventions as described above.
    * A highly effective method of contraception is defined as one that results in a low failure rate (less than 1% per year) when used consistently and correctly. Note that some contraception methods are not considered highly effective. The participants chosen method(s) must be confirmed as highly effective prior to study entry.
12. Participant is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants must not meet any of the following criteria:

1. Have locally confirmed DNA-mismatch repair deficient or microsatellite instability (MSI) status - high Stage IV colorectal cancer.
2. Participants with brain metastases may participate provided they are clinically stable for at least 4 weeks prior to study entry, have no evidence of new or enlarging brain metastases and are off steroids for at least 7 days.
3. Have a concurrent malignancy or have had another malignancy within the past 5 years prior to screening that is expected to alter life expectancy or may interfere with disease assessment.
4. Have Type 1 or 2 diabetes mellitus.
5. Have Reversible Posterior Leukoencephalopathy.
6. Have a history of or evidence of active gastrointestinal perforation or gastrointestinal fistula.
7. Have a family history of a genetic / familial neuropathy.
8. Have pre-existing clinical neuropathy ≥ Grade 2 per CTCAE v5.0 from any cause.
9. Have had major surgery other than a minor outpatient procedure within 28 days prior to randomization or have not recovered from major side effects of the surgery if more than 4 weeks have elapsed since surgery.
10. Have poorly controlled hypertension despite the use of antihypertensive agents defined as blood pressure > 150/90 mmHg on at least 2 repeated determinations on separate days during screening period.
11. Have a history of cardiac dysfunction including:

    * Myocardial infarction within 6 months prior to initiation of screening.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV) within 6 months prior to initiation of screening
    * Active cardiomyopathy.
    * Electrocardiogram with QTc > 470 milliseconds at screening.
12. Have uncontrolled severe infections (acute or chronic) including HIV, Hepatitis B or C
13. Have active poor wound healing (delayed healing, wound infection or fistula).
14. Have evidence of active, clinically significant bleeding (e.g., gastrointestinal bleeding, hemoptysis, or gross hematuria) at screening. No bleeding diathesis, hemorrhage, or arterial/ venous thrombotic events within 6 months prior to initiation of screening, including transient ischemic attack, cerebrovascular accident, unstable angina or angina requiring surgical or medical intervention in the past 6 months, or myocardial infarction. Patients with clinically significant peripheral artery disease (i.e., claudication on less than one block) or any other arterial thrombotic event are also ineligible.
15. Are breast feeding or pregnant, confirmed by a positive serum human chorionic gonadotropin (hCG) laboratory test.
16. Have other concurrent severe and/or uncontrolled medical condition that would, in the Investigator's judgment contraindicate the participant's participation in the clinical study or obscure proper assessment of safety and toxicity of the prescribed regimen.
17. Have received prior treatment with any investigational drug within 4 weeks (28 days) prior to randomization.
18. Have received prior treatment with neurotoxic chemotherapy including but not limited to oxaliplatin, cisplatin, a taxane, or a vinca alkaloid.
19. Have received prior treatment with any anti-VEGF agent.
20. Are receiving any agent for the treatment, prevention, or with known/hypothesized efficacy for peripheral neuropathy; including but not limited to gabapentin, pregabalin, venlafaxine, duloxetine, amitriptyline, nortriptyline, or anti-neuropathic pain topical cream.
21. Have a known sensitivity to the components of BXQ-350 (SapC and DOPS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose | 6 months
  To determine the recommended phase 2 dose of BXQ-350, when given with mFOLFOX7 and bevacizumab, according to the investigational product (IP) related dose limiting toxicities (DLTs).
Incidence of Treatment Emergent Adverse Events as Assessed by CTCAE v5.0 | 6 months
  To determine the safety of BXQ-350 when given with mFOLFOX7 and bevacizumab, as evidenced by the incidence of treatment emergent adverse events assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Objective Response Rate (ORR) | 6 months
  To determine the ORR of BXQ-350 when given with mFOLFOX7 and bevacizumab. ORR is defined as the percentage of participants with evidence of a complete or partial response as per the Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 6 months
  To evaluate the Cmax of BXQ-350 in combination with mFOLFOX7 and bevacizumab.
Overall Survival (OS) | 6 months
  To evaluate OS in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab. OS is defined as the time from the date of randomization until date of death due to any cause.
Progression Free Survival (PFS) | 6 months
  To evaluate PFS in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab. PFS is defined as the time from the date of randomization until date of disease progression or death.
Duration of Response (DoR) | 6 months
  To evaluate DoR in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab. DoR is defined as the time from documentation of disease response to disease progression according to RECIST.
Disease Control Rate (DCR) | 6 months
  To evaluate DCR in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab. DCR is defined as the proportion of participants whose best overall response (BOR) was complete (CR), partial response (PR) and stable disease (SD) according to RECIST.
Total Sensory Neuropathy | 6 months
  To evaluate chronic neuropathy symptoms in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab. Total sensory neuropathy scores will be obtained from the EORTC QLQ-CIPN20 questionnaire.
CIPN Assessment | 6 months
  To evaluate acute CIPN symptoms in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab utilizing the CIPN Assessment Tool questionnaire.
Post Oxaliplatin Assessment | 6 months
  To evaluate acute CIPN symptoms post oxaliplatin dosing in participants receiving BXQ-350 with mFOLFOX7 and bevacizumab utilizing the Post-oxaliplatin Symptom questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Study Director — Bexion Pharmaceuticals, Inc.
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UC Irvine Health, Orange, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Sylvester Comprehensive Cancer Center, University of Miami Hospitals and Clinics, Miami, Florida
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Louisville, James Graham Brown Cancer Center, Louisville, Kentucky
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Stony Brook Cancer Center, Stony Brook, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio